CLINICAL TRIAL: NCT05157945
Title: AN OPEN-LABEL STUDY OF ALTO-300 IN ADULTS WITH MAJOR DEPRESSIVE DISORDER
Brief Title: ALTO-300 in Depression (ALTO-300-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTO-300-004
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTO-300 (Experimental): ALTO-300 tablet PO; daily dosing 8 weeks
  Interventions: Drug: ALTO-300 PO Tablet

INTERVENTIONS:
Drug: ALTO-300 PO Tablet — One tablet daily

SUMMARY:
The purpose of this study is to collect biologically-based data for defining predictors and correlates of the effects of ALTO-300.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate to severe major depressive disorder
* Currently taking a SSRI, SNRI, or bupropion for at least 6 weeks with no dose modifications in the past 2 weeks
* Must have failed to adequately respond to the current antidepressant medication
* Willing to comply with all study assessments and procedures
* Must not be pregnant or breastfeeding at time of enrollment or throughout study

Exclusion Criteria:

* Evidence of liver impairment or disease
* Active suicidal ideation
* Moderate to severe Alcohol Use Disorder
* Diagnosed bipolar disorder or psychotic disorder
* Has a history of hypersensitivity or allergic reaction to ALTO-300 or any of its components/excipients
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
To understand the relationship between baseline biology and change in the Montgomery-Asberg Depression Rating Scale (MADRS) with ALTO-300 | Measured 6 times over 8 weeks
  The Montgomery-Åsberg Depression Rating Scale (MADRS) measures the severity of depression where smaller scores indicate less depression and higher scores suggest more severe depression. Possible scores for this 10 item version range from 0 to 60. The change from baseline to the end of the study is the primary outcome.
To understand the relationship between baseline biology and change in the Clinical Global Impression scale - Severity (CGI-S) with ALTO-300 | Measured 6 times over 8 weeks
  The Clinical Global Impression scale - Severity (CGI-S) measures the severity of psychopathology in general where smaller scores indicate less illness and higher scores suggest more severe illness. Possible scores for this scale range from 1 to 7. The change from baseline to the end of the study is the primary outcome.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability of ALTO-300 | From the signing of the ICF until the follow-up visit (up to 12 weeks)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants With Clinically Significant Vital Signs Abnormalities as a Measure of Safety and Tolerability of ALTO-300 | From the signing of the ICF until the end-of-treatment visit (up to 11 weeks)]
  Vital signs measured include blood pressure, heart rate, respiratory rate, temperature, and weight.
Number of Participants With Clinically Significant Laboratory Abnormalities as a Measure of Safety and Tolerability of ALTO-300 | From the signing of the ICF until the end-of-treatment visit (up to 11 weeks)]
  Blood samples for serum chemistry and hematology will be collected for clinical laboratory testing.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cerebral - Atlanta, Atlanta, Georgia
  - Site 171, Jackson, Mississippi
  - Cerebral - New York City, New York, New York
  - Cerebral - Dallas, Dallas, Texas